CLINICAL TRIAL: NCT05148637
Title: The Effect of Different Modalities of General Anesthesia and Regional Cerebral Oxygenation on Postoperative Cognitive Dysfunction in Elderly Patients Undergoing Spine Surgery in Prone Position
Brief Title: General Anesthesia and Regional Cerebral Oxygenation inSpine Surgery Prone Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Mogahed, Associate professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 34775/7/21
Record Dates: First submitted 2021-10-29; First posted 2021-12-08 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Spinal Disease
MeSH Terms: conditions — Spinal Diseases | interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Intervention Model Description: Montreal Cognitive Assessment (MoCA) were used to assess cognitive function the day before surgery and seventh postoperative day.
Who Masked: Participant
Masking Description: The methods of anesthesia were described to the enrolled patients preoperatively, but the patients were unaware about their group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Active Comparator): anesthesia maintained by sevoflurane
  Interventions: Drug: Maintenance of general anesthesia by Sevoflurane
- Group II (Active Comparator): anesthesia maintained by desflurane
  Interventions: Drug: Maintenance of general anesthesia by Desflurane
- Group III (Active Comparator): anesthesia maintained by TIVA
  Interventions: Drug: Anesthesia was maintained by inhalational anesthesia (total intravenous anesthesia by lidocaine, propfol and fentanyl infusions)

INTERVENTIONS:
Drug: Maintenance of general anesthesia by Sevoflurane — Anesthesia was maintained by inhalational anesthesia (sevoflurane) titrated by monitoring of patient sensitivity index of the Masimo
  Other Names: Sevoflurane
  Arms: Group I
Drug: Maintenance of general anesthesia by Desflurane — Anesthesia was maintained by inhalational anesthesia (desflurane) titrated by monitoring of patient sensitivity index of the Masimo
  Other Names: Desflurane
  Arms: Group II
Drug: Anesthesia was maintained by inhalational anesthesia (total intravenous anesthesia by lidocaine, propfol and fentanyl infusions) — Anesthesia was maintained by inhalational anesthesia (total intravenous anesthesia by lidocaine, propfol and fentanyl infusions) titrated by monitoring of patient sensitivity index of the Masimo
  Other Names: Total intravenous anesthesia
  Arms: Group III

SUMMARY:
Elderly patients are reportedly at higher risk of postoperative cognitive dysfunction (POCD).The authors hypothesized that the incidence of POCD would be affected by several factors including, the age of the patient, the degree of cerebral oxygenation, type of anesthesia administered, majority of surgery and the patient position during surgery.The investigators examined the relationship between all the previous parameters and (POCD).

DETAILED DESCRIPTION:
105 patients 65 years or older and scheduled for lumbar spinal surgery will be enrolled. Enrolled patients have either degenerative lumbar spinal stenosis or spinal cord tumor. The planned surgical procedures will be all performed in the prone position using the Wilson frame with the head and neck in the neutral position and included laminectomy and discectomy, spinal fusion, and (when present) removal of the spinal cord tumor. Written informed consent for participation in this study will be obtained from all patients.

Patients will be screened within 1 week before the scheduled surgery. Details and medical comorbidities, Inclusion criteria were as follows: elective spine surgery in prone position, 60-75 years old, American Society of Anesthesiologists (ASA) physical status score of I,II or III, and body mass index (BMI) ranging from 22 to 45 kg/m2 , patients should have a sufficient level of education to be capable of completing neuropsychological tests; a pre-operative mini mental state examination (MMSE) score ≥23. Exclusion criteria were as follows: preexisting neuropsychiatric disorders or inability to correctly perform neurocognitive tests on the patient, emergency operation, diagnosis of coma, depression, cognitive impairment, cardiovascular, respiratory or central nervous system disease, renal or hepatic dysfunction or serious hearing or visual impairment;

In the operating room, Patients were monitored by 5 lead electrocardiogram, invasive arterial blood pressure (IABP) through the arterial catheter and (Masimo®, Irvine, CA) which provides non-invasive continuous technologies for monitoring and measuring many physiological variables such as arterial oxygen saturation (SpO2), heart rate (HR) and hemoglobin concentration (Hb%), end tidal CO2, noninvasive blood pressure, body temperature, (O3 ®, Masimo, Irvine, CA) attached to the patient to provide continuous monitoring of regional cerebral oxygen saturation (rSO2) of the two sides by a near-infrared spectroscopy sensors. (SedLine ®, Masimo, CA) brain function monitoring by Patient State Index (PSI) which is a processed EEG parameter affected by the anesthetic agents.

Patients were randomly divided into three groups 35 each; group I: anesthesia maintained by sevoflurane, group II: anesthesia maintained by desflurane, and group III: anesthesia maintained by TIVA. In all groups the doses of anesthetics were adjusted to maintain (Psi) (patient sensitivity index) between 25-50% measured by (SedLine, Masimo®, CA) rocuronium boluses were given to maintain stable neuromuscular block.

Anesthesia was managed according to a standardized protocol that was identical for each group. Following 3 min of pre-oxygenation (with 100 % O2), anesthesia was induced by slow intravenous injection of propofol (1-2 mg/kg), fentanil (1-μg /kg). Tracheal intubation was facilitated with Rocrunium (0.4-0.6mg/kg) Mechanical ventilation was initiated with a tidal volume of 7 ml/kg, a respiratory rate of 12 /min, a positive end expiratory pressure of 5 cmH2O and inspiratory-expiratory ratio of 1:2 to maintain PETCO2 in the range 35-40 mmHg. Oxygen flow rate was set at 2 l/min.

Anesthesia was maintained in the three Groups by sevoflurane , desflurane, and propofol to target PSI to 25-50 fentanyl 100μg/h and boluses of rocrunium were used to supplement maintenance of anesthesia.

Patients' demographic and basic clinical characteristics, fluid balance, blood loss, duration of surgery, temperature, time taken for recovery of spontaneous breathing, eye opening on command and time taken for extubation were also recorded. HR, mean arterial pressure (MAP) and central venous pressure were recorded at five perioperative time points: on entering the operating room (T0); before tracheal intubation (T1); before surgery (T2); immediately after surgery (T3) and immediately after tracheal extubation (T4). . In the operating room, patients were laid in the supine position, and a The patient's baseline rSO2 data were acquired before anesthetic induction while the patient breathed room air. The anesthesiologists and surgeons were blinded to the rSO2 data, which wererecorded at 30-second intervals on the device's accessory disk drive for later analysis. No interventions were attempted based on the device. Both the right and the left frontal rSO2 values wererecorded simultaneously, and the lower value of either side werecollected for analysis.

Assessment of perioperative cognitive function The MMSE and Montreal Cognitive Assessment (MoCA) were used to assess cognitive function the day before surgery and seventh postoperative day. All data collectors had undergone standard training, and were blinded to the randomization status of the participants. The MMSE consists of tests of orientation (in time and place), memory (immediate and short-term), calculation, language (naming, repetition, listening and reading comprehension, writing), visual spatial awareness, concentration and attention, and is suitable for detecting more severe cognitive dysfunction. The MoCA tests visuospatial and executive function (alternate trail making test, copy the cube, clock drawing), language ability, attention and calculation, delayed recall and abstract thinking, and can detect milder cognitive dysfunction. Patients' cognitive function was evaluated by MoCA if the MMSE score equaled or exceeded 23.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for lumbar spinal surgery
* Procedures performed in the prone position

Exclusion Criteria:

* preexisting neuropsychiatric disorders
* emergency operation
* cardiovascular disease
* respiratory disease
* central nervous system disease
* renal dysfunction
* hepatic dysfunction

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Assessment of postoperative cognitive function | 7 days
  Assessment of postoperative cognitive function using mini mental state examination to assess patient's orientation postoperatively by 30-point questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Mona Mohamed Mogahed, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes